CLINICAL TRIAL: NCT02937701
Title: A Randomized, Double-Blind Phase 3 Study to Assess the Efficacy and Safety of ABP 710 Compared to Infliximab in Subjects With Moderate to Severe Rheumatoid Arthritis
Brief Title: Study to Assess if ABP710 is Safe & Effective in Treating Moderate to Severe Rheumatoid Arthritis Compared to Infliximab
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Amgen (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 20140111; 2014-004704-29 (EudraCT Number)
Record Dates: First submitted 2016-08-30; First posted 2016-10-19 (Estimated); Results first posted 2019-08-28 (Actual); Last update posted 2019-08-28 (Actual); Status verified 2019-08

CONDITIONS: Arthritis, Rheumatoid
MeSH Terms: conditions — Arthritis, Rheumatoid | interventions — Infliximab

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- ABP 710 (Experimental): Participants randomized to receive a 3 mg/kg intravenous (IV) infusion of ABP 710 on day 1, at weeks 2 and 6, and every 8 weeks thereafter until week 22.
  At week 22 participants continued receiving 3 mg/kg ABP 710 every 8 weeks through week 46.
  Interventions: Biological: ABP 710
- Infliximab (Active Comparator): Participants randomized to receive a 3 mg/kg IV infusion of infliximab on day 1, at weeks 2 and 6, and every 8 weeks thereafter until week 22.
  At week 22 participants were re-randomized in a 1:1 ratio to either continue receiving 3 mg/kg infliximab every 8 weeks or transition to receive 3 mg/kg ABP 710 every 8 weeks through week 46.
  Interventions: Biological: Infliximab

INTERVENTIONS:
Biological: ABP 710 — Administered by intravenous infusion
  Arms: ABP 710
Biological: Infliximab — Administered by intravenous infusion
  Other Names: Remicade®
  Arms: Infliximab

SUMMARY:
The main purpose of the study was to compare rheumatoid arthritis symptom improvement in participants who were given ABP 710 to those who were given infliximab, 22 weeks after starting treatment.

ELIGIBILITY:
Inclusion Criteria:

* Subject (man or woman) is ≥ 18 and ≤ 80 years old.
* Subject is diagnosed with rheumatoid arthritis (RA) as determined by meeting the 2010 American College of Rheumatology (ACR)/European League Against Rheumatism classification criteria for RA.
* Subject has RA duration of at least 3 months.
* Subject has active RA defined as ≥ 6 swollen joints and ≥ 6 tender joints (based on 66/68 joint count excluding distal interphalangeal joints) at screening and baseline and at least 1 of the following at screening:

  * erythrocyte sedimentation rate ≥ 28 mm/hr
  * serum C-reactive protein > 1.0 mg/dL
* Subject has a positive rheumatoid factor or anti-cyclic citrullinated peptide at screening.
* Subject has taken methotrexate (MTX) for ≥ 12 consecutive weeks and is on a stable dose of oral or subcutaneous MTX 7.5 to 25 mg/week for ≥ 8 weeks before receiving the investigational product and is willing to remain on a stable dose throughout the study.
* For a subject on nonsteroidal anti-inflammatory drugs (NSAIDs) or low potency analgesics such as tramadol, Soma Compounds, Fioricet, or Fiorinal, the dose should be stable for ≥ 2 weeks before screening.
* For a subject on oral corticosteroids (≤ 10 mg prednisone or equivalent), the dose should be stable for ≥ 4 weeks before screening.
* Subject has no known history of active tuberculosis.
* Subject has a negative test for tuberculosis during screening defined as either:

  * negative purified protein derivative (PPD) defined as < 5 mm of induration at 48 to 72 hours after test is placed OR
  * negative Quantiferon test
* Subject with a positive PPD and a history of Bacillus Calmette-Guérin vaccination is allowed with a negative Quantiferon test.
* Subject with a positive PPD test (without a history of Bacillus Calmette-Guérin vaccination) or a subject with a positive or indeterminate Quantiferon test is allowed if they have all of the following:

  * no symptoms of tuberculosis according to the worksheet provided by the sponsor, Amgen Inc.
  * documented history of adequate prophylaxis initiation before receiving investigational product in accordance with local recommendations
  * no known exposure to a case of active tuberculosis after most recent prophylaxis

Exclusion Criteria:

* Subject has a history of prosthetic or native joint infection.
* Subject has an active infection or history of infections as follows:

  * any active infection for which systemic anti-infectives were used within 28 days before first dose of investigational product
  * a serious infection, defined as requiring hospitalization or intravenous (IV) anti-infective(s) within 8 weeks before the first dose of investigational product
  * recurrent or chronic infections or other active infection that, in the opinion of the investigator, might cause this study to be detrimental to the subject
* Subject has a positive blood test for human immunodeficiency virus (HIV).
* Subject has a positive hepatitis B surface antigen, hepatitis B core antibody, or hepatitis C virus antibody result at screening.
* Subject has uncontrolled, clinically significant systemic disease such as diabetes mellitus, cardiovascular disease including moderate or severe heart failure (New York Heart Association Class III/IV), renal disease, liver disease, or hypertension.
* Subject had a malignancy within 5 years EXCEPT for treated and considered cured cutaneous squamous or basal cell carcinoma, in situ cervical cancer, OR in situ breast ductal carcinoma.
* Subject has a history of neurologic symptoms suggestive of central or peripheral nervous system demyelinating disease.
* Subject has a major chronic inflammatory disease or connective tissue disease other than RA, with the exception of secondary Sjögren's syndrome.
* Subject has a concurrent medical condition that, in the opinion of the investigator, could cause this study to be detrimental to the subject.
* Subject has laboratory abnormalities at screening, including any of the following:

  * hemoglobin < 9 g/dL
  * platelet count < 100 000/mm³
  * white blood cell count < 3 000/mm³
  * aspartate aminotransferase and/or alanine aminotransferase ≥ 2.0 x the upper limit of normal
  * creatinine clearance < 50 mL/min (Cockroft-Gault formula)
  * any other laboratory abnormality, that, in the opinion of the investigator, will prevent the subject from completing the study or will interfere with the interpretation of the study results.
* Subject has used commercially available or investigational biologic therapies for RA as follows:

  * anakinra, etanercept within 1 month before the first dose of investigational product
  * abatacept, tocilizumab, adalimumab, golimumab, certolizumab within 3 months before the first dose of investigational product
  * other experimental or commercially available biologic therapies for RA within 3 months or 5 half-lives (whichever is longer) before the first dose of investigational product
  * rituximab within 9 months before the investigational product along with evidence of incomplete B cell recovery
* Subject has received live vaccines within 28 days before the first dose of investigational product or plans to receive live vaccines during the course of the study.
* Subject has previously received Remicade® (infliximab) or a biosimilar of infliximab.
* Woman who is pregnant or breast feeding, or plans to become pregnant while enrolled in the study and for 6 months after the last dose of investigational product.
* Women of childbearing potential (ie, neither surgically sterile nor postmenopausal) and do not agree to use adequate contraception (eg, true abstinence, sterilization, birth control pills, Depo-Provera® [medroxyprogesterone] injections, or contraceptive implants) while on study and for 6 months after the last dose of investigational product.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 558 (Actual)
Dates: Start 2016-10-10 (Actual); Primary Completion 2018-04-16 (Actual); Study Completion 2018-08-13 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: MD, Study Director — Amgen
Locations (66):
- United States (26):
  - Research Site, Huntsville, Alabama
  - Research Site, Tuscaloosa, Alabama
  - Research Site, Peoria, Arizona
  - Research Site, Covina, California
  - Research Site, Hemet, California
  - Research Site, Upland, California
  - Research Site, Van Nuys, California
  - Research Site, Aventura, Florida
  - Research Site, Miami Lakes, Florida
  - Research Site, Orlando, Florida
  - Research Site, Sarasota, Florida
  - Research Site, Vero Beach, Florida
  - Research Site, Lexington, Kentucky
  - Research Site, Grand Blanc, Michigan
  - Research Site, Flowood, Mississippi
  - Research Site, St Louis, Missouri
  - Research Site, Omaha, Nebraska
  - Research Site, Voorhees Township, New Jersey
  - Research Site, Charlotte, North Carolina
  - Research Site, Charleston, South Carolina
  - Research Site, Memphis, Tennessee
  - Research Site, Carrollton, Texas
  - Research Site, Dallas, Texas
  - Research Site, Houston, Texas
  - Research Site, League City, Texas
  - Research Site, Plano, Texas
- Australia (2):
  - Research Site, Woodville, South Australia
  - Research Site, Fitzroy, Victoria
- Bulgaria (5):
  - Research Site, Sofia, Sofia
  - Research Site, Pleven
  - Research Site, Plovdiv
  - Research Site, Sliven
  - Research Site, Varna
- Canada (2):
  - Research Site, Victoria, British Columbia
  - Research Site, Saint Johns, Newfoundland and Labrador
- Czechia (7):
  - Research Site, Brno, Jihormoravsky KRAJ
  - Research Site, Hlučín, Moravskoslezský kraj
  - Research Site, Prague, Prague
  - Research Site, Liberec, Severocesky KRAJ
  - Research Site, Ostrava, Severomoravsky KRAJ
  - Research Site, Zlín, Severomoravsky KRAJ
  - Research Site, Pardubice, Vychodocesky KRAJ
- Germany (4):
  - Research Site, Hildesheim, Lower Saxony
  - Research Site, Bad Doberan, Mecklenburg-Vorpommern
  - Research Site, Magdeburg, Saxony-Anhalt
  - Research Site, Hamburg
- Hungary (4):
  - Research Site, Gyula, Bekes County
  - Research Site, Szentes, Csongrád megye
  - Research Site, Győr, Győr-Moson-Sopron
  - Research Site, Veszprém, Veszprém megye
- Poland (13):
  - Research Site, Poznan, Greater Poland Voivodeship
  - Research Site, Bydgoszcz, Kuyavian-Pomeranian Voivodeship
  - Research Site, Torun, Kuyavian-Pomeranian Voivodeship
  - Research Site, Krakow, Lesser Poland Voivodeship
  - Research Site, Wroclaw, Lower Silesian Voivodeship
  - Research Site, Lublin, Lublin Voivodeship
  - Research Site, Warsaw, Masovian Voivodeship
  - Research Site, Stalowa Wola, Podkarpackie Voivodeship
  - Research Site, Bialystok, Podlaskie Voivodeship
  - Research Site, Gdansk, Pomeranian Voivodeship
  - Research Site, Katowice, Silesian Voivodeship
  - Research Site, Elblag, Warmian-Masurian Voivodeship
  - Research Site, Lodz, Łódź Voivodeship
- Spain (3):
  - Research Site, Barcelona
  - Research Site, Madrid
  - Research Site, Seville

REFERENCES:
- [Derived] Genovese MC, Sanchez-Burson J, Oh M, Balazs E, Neal J, Everding A, Hala T, Wojciechowski R, Fanjiang G, Cohen S. Comparative clinical efficacy and safety of the proposed biosimilar ABP 710 with infliximab reference product in patients with rheumatoid arthritis. Arthritis Res Ther. 2020 Mar 26;22(1):60. doi: 10.1186/s13075-020-2142-1. PMID 32216829
- See also: AmgenTrials clinical trials website — http://www.amgentrials.com

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This study was conducted at 75 centers in Australia, Bulgaria, Canada, Czech Republic, Germany, Hungary, Poland, Spain, and the United States.
Pre-assignment Details: Participants were randomized in a 1:1 ratio to receive ABP 710 or infliximab, stratified by geographic region and prior biologic use.
  At week 22 participants initially randomized to infliximab were re-randomized in a 1:1 ratio to continue infliximab or switch to ABP 710. Participants initially randomized to ABP 710 continued receiving ABP 710.
Groups:
- ABP 710: Participants randomized to receive a 3 mg/kg intravenous (IV) infusion of ABP 710 on day 1, at weeks 2 and 6, and every 8 weeks thereafter until week 22.
- Infliximab: Participants randomized to receive 3 mg/kg IV infusion of infliximab on day 1, at weeks 2 and 6, and every 8 weeks thereafter until week 22.
- ABP 710 / ABP 710: At week 22 participants initially randomized to ABP 710 continued receiving 3 mg/kg ABP 710 every 8 weeks through week 46.
- Infliximab / Infliximab: At week 22 participants initially randomized to infliximab were re-randomized to continue receiving 3 mg/kg infliximab every 8 weeks through week 46.
- Infliximab / ABP 710: At week 22 participants initially randomized to infliximab were re-randomized to receive 3 mg/kg ABP 710 every 8 weeks through week 46.
Period: Day 1 to Week 22
Arm/Group | ABP 710 | Infliximab | ABP 710 / ABP 710 | Infliximab / Infliximab | Infliximab / ABP 710
Started | 279 | 279 | 0 | 0 | 0
Received Treatment | 278 | 278 | 0 | 0 | 0
Completed | 244 | 240 | 0 | 0 | 0
Not Completed | 35 | 39 | 0 | 0 | 0
Not completed — Adverse Event | 11 | 14 | 0 | 0 | 0
Not completed — Protocol Specified Criteria | 7 | 7 | 0 | 0 | 0
Not completed — Dissatisfied With Treatment Efficacy | 5 | 9 | 0 | 0 | 0
Not completed — Withdrawal by Subject | 6 | 6 | 0 | 0 | 0
Not completed — Death | 1 | 1 | 0 | 0 | 0
Not completed — Protocol Violation | 1 | 1 | 0 | 0 | 0
Not completed — Lost to Follow-up | 1 | 1 | 0 | 0 | 0
Not completed — Physician Decision | 2 | 0 | 0 | 0 | 0
Not completed — Other | 1 | 0 | 0 | 0 | 0
Period: Week 22 to Week 50
Arm/Group | ABP 710 | Infliximab | ABP 710 / ABP 710 | Infliximab / Infliximab | Infliximab / ABP 710
Started | 0 | 0 | 244 | 121 | 119
Completed | 0 | 0 | 212 | 113 | 110
Not Completed | 0 | 0 | 32 | 8 | 9
Not completed — Adverse Event | 0 | 0 | 10 | 3 | 3
Not completed — Dissatisfied with Treatment Efficacy | 0 | 0 | 10 | 3 | 2
Not completed — Withdrawal by Subject | 0 | 0 | 8 | 2 | 1
Not completed — Lost to Follow-up | 0 | 0 | 2 | 0 | 1
Not completed — Physician Decision | 0 | 0 | 2 | 0 | 1
Not completed — Other | 0 | 0 | 0 | 0 | 1

BASELINE CHARACTERISTICS:
Population: The intent-to-treat analysis set included all randomized participants
Groups:
- Total: Total of all reporting groups
Arm/Group | ABP 710 | Infliximab | Total
Number analyzed (Participants) | 279 | 279 | 558
Age, Continuous [Mean (Standard Deviation); unit: years] | 55.0 (11.72) | 54.8 (11.42) | 54.9 (11.56)
Age, Customized [Count of Participants; unit: Participants]
  < 65 years | 217 | 217 | 434
  ≥ 65 years | 62 | 62 | 124
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 214 | 223 | 437
  Male | 65 | 56 | 121
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 18 | 13 | 31
  Not Hispanic or Latino | 261 | 266 | 527
  Unknown or Not Reported | 0 | 0 | 0
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  White | 265 | 267 | 532
  Black or African American | 12 | 12 | 24
  Asian | 2 | 0 | 2
Geographic Region [Count of Participants; unit: Participants]
  Asia Pacific | 5 | 4 | 9
  Europe | 220 | 222 | 442
  North America | 54 | 53 | 107
Prior Biologic Use for Rheumatoid Arthritis [Count of Participants; unit: Participants]
  Yes | 77 | 81 | 158
  No | 202 | 198 | 400
Duration of Rheumatoid Arthritis (RA) [Mean (Standard Deviation); unit: years] | 8.72 (7.914) | 8.34 (7.604) | 8.53 (7.756)
Swollen joint Count [Mean (Standard Deviation); unit: joints] — A total of 66 joints were scored for presence or absence of swelling.
  joints | 14.595 (8.0507) | 14.730 (8.8315) | 14.663 (8.4428)
Tender Joint Count [Mean (Standard Deviation); unit: joints] — A total of 68 joints were scored for presence or absence of tenderness.
  joints | 23.109 (12.1648) | 23.764 (13.3800) | 23.436 (12.7796)
Patient Global Health Assessment [Mean (Standard Deviation); unit: mm] — The participant's overall assessment of their disease activity in the past week assessed on a 100 mm visual analog scale (VAS), where 0 mm = No RA activity at all and 100 mm = Worst RA activity imaginable. Population: Participants with available data
  mm
    number analyzed (Participants) | 278 | 278 | 556
    (all) | 65.4 (18.13) | 64.1 (20.03) | 64.7 (19.10)
Investigator's Global Health Assessment [Mean (Standard Deviation); unit: mm] — The investigator's assessment of the participant's current disease activity assessed on a 100 mm VAS where 0 mm = no activity at all (symptom-free and no arthritis symptoms) and 100 mm = worst activity imaginable (maximum arthritis disease activity). Population: Participants with available data
  mm
    number analyzed (Participants) | 278 | 278 | 556
    (all) | 64.5 (15.88) | 64.1 (15.76) | 64.3 (15.81)
Patient's Assessment of Disease-related Pain [Mean (Standard Deviation); unit: mm] — The participant's assessment of their current level of pain assessed on a 100 mm horizontal VAS, where 0 mm = no pain at all and 100 mm = worst pain imaginable.
  mm | 63.5 (20.30) | 61.5 (21.65) | 62.5 (20.99)
Disability Index of the Health Assessment Questionnaire (HAQ-DI) [Mean (Standard Deviation); unit: units on a scale] — The HAQ-DI is a patient-reported questionnaire consisting of 20 questions in eight domains: dressing/grooming, arising, eating, walking, hygiene, reach, grip, and usual activities. Participants assessed their ability to do each task over the past week using the following response categories: without any difficulty (0); with some difficulty (1); with much difficulty (2); and unable to do (3). Scores on each task are summed and averaged to provide an overall score ranging from 0 to 3, where zero represents no disability and three very severe, high-dependency disability. Population: Participants with available data
  units on a scale
    number analyzed (Participants) | 278 | 278 | 556
    (all) | 1.44 (0.584) | 1.42 (0.617) | 1.43 (0.601)
C-reactive Protein (CRP) Concentration [Mean (Standard Deviation); unit: mg/L] — C-reactive protein (CRP) is a protein found in blood. CRP levels rise in response to inflammation.
  mg/L | 14.26 (20.171) | 14.64 (23.117) | 14.45 (21.675)

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants With an American College of Rheumatology 20% (ACR20) Response at Week 22
Description: The primary efficacy endpoint was the response difference (RD) of 20% improvement in ACR core set measurements (ACR20) at week 22.
  A positive ACR20 response is defined if the following 3 criteria for improvement from baseline were met:
  * ≥ 20% improvement in 68 tender joint count;
  * ≥ 20% improvement in 66 swollen joint count; and
  * ≥ 20% improvement in at least 3 of the 5 following parameters:
    * Patient's assessment of disease-related pain (measured on a 100 mm visual analog scale [VAS]);
    * Patient's global health assessment (measured on a 100 mm VAS);
    * Investigator's global health assessment (measured on a 100 mm VAS);
    * Patient's self-assessment of physical function (Health Assessment Questionnaire - Disability Index [HAQ-DI]);
    * C-reactive protein concentration.
Time Frame: Baseline and week 22
Population: Intent-to-treat population; Participants with missing data at week 22 were counted as non-responders
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | ABP 710 | Infliximab
Number analyzed (Participants) | 279 | 279
percentage of participants | 68.1 [62.63 to 73.57] | 59.1 [53.37 to 64.91]
Statistical Analysis 1: Comparison: ABP 710 vs Infliximab; For the primary analysis of ACR20, the response difference (RD) was estimated by the Mantel-Haenszel (MH) estimate and the 90% confidence intervals (CIs) of RD were estimated from the stratified Newcombe confidence limits, adjusting for actual stratification factors (geographic region and prior biologic use for RA); Test type: Equivalence — Clinical equivalence for the primary endpoint was to be evaluated sequentially by first comparing the 2-sided 90% CI for RD of ACR20 at week 22 between ABP 710 and infliximab with an equivalence margin of (-15%, 15%). If the first test was successful, RD of ACR20 at week 22 was to be further evaluated by comparing the 2-sided 90% CI between ABP 710 and infliximab with an equivalence margin of (-12%, 15%); Response Difference = 9.37, 90% CI 2-sided [2.67 to 15.96]
Statistical Analysis 2: Comparison: ABP 710 vs Infliximab; A sensitivity analysis with the RD estimate and CIs for RD of ACR20 estimated using a generalized linear model with geographic region and prior biologic use for RA as covariates was also conducted; Test type: Equivalence — [test comment as in outcome 1, analysis 1]; Response Difference = 9.30, 90% CI 2-sided [2.67 to 15.92] — Response Difference is based on a generalized linear model with actual stratification variables (geographic region and prior biologic use for RA) as covariates in the model
Statistical Analysis 3: Comparison: ABP 710 vs Infliximab; A post-hoc analysis was conducted to adjust for the impact of random imbalance in baseline demographic and disease characteristics between the 2 treatment groups. The MH estimate of RD and corresponding CIs were estimated using a nonparametric analysis of covariance method with stratification factors geographic region and prior biologic use, and adjustment for baseline covariates (ACR core set, age, use of oral corticosteroid, use of NSAID, body mass index categories, and methotrexate dose); Test type: Equivalence — [test comment as in outcome 1, analysis 1]; Response Difference = 7.184, 90% CI 2-sided [0.748 to 13.620] — The ACR core set includes tender joint count, swollen joint count, subject's global health assessment, investigator's global health assessment, subject's assessment of disease related pain, HAQ-DI, and CRP

2. Secondary Outcome: Percentage of Participants With an ACR20 Response Through Week 14
Description: A positive ACR20 response is defined if the following 3 criteria for improvement from baseline were met:
  * ≥ 20% improvement in 68 tender joint count;
  * ≥ 20% improvement in 66 swollen joint count; and
  * ≥ 20% improvement in at least 3 of the 5 following parameters:
    * Patient's assessment of disease-related pain (measured on a 100 mm visual analog scale [VAS]);
    * Patient's global health assessment (measured on a 100 mm VAS);
    * Investigator's global health assessment (measured on a 100 mm VAS);
    * Patient's self-assessment of physical function (Health Assessment Questionnaire - Disability Index [HAQ-DI]);
    * C-reactive protein concentration.
Time Frame: Baseline and weeks 2, 6, and 14
Population: Intent-to-treat population; participants with missing data at a given visit were counted as non-responders.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | ABP 710 | Infliximab
Number analyzed (Participants) | 279 | 279
percentage of participants
  Week 2 | 46.2 [40.39 to 52.09] | 38.0 [32.30 to 43.69]
  Week 6 | 64.9 [59.27 to 70.48] | 59.9 [54.10 to 65.61]
  Week 14 | 66.3 [60.76 to 71.85] | 60.2 [54.47 to 65.96]
Statistical Analysis 1: Comparison: ABP 710 vs Infliximab; The response difference at week 2 was estimated by the Mantel-Haenszel estimate; 90% confidence intervals were estimated from the stratified Newcombe confidence limits, adjusting for actual stratification factors (geographic region and prior biologic use); Test type: Other; Response Difference = 8.03, 90% CI 2-sided [1.15 to 14.81]
Statistical Analysis 2: Comparison: ABP 710 vs Infliximab; The response difference at week 6 was estimated by the Mantel-Haenszel estimate; 90% confidence intervals were estimated from the stratified Newcombe confidence limits, adjusting for actual stratification factors (geographic region and prior biologic use); Test type: Other; Response Difference = 4.96, 90% CI 2-sided [-1.80 to 11.64]
Statistical Analysis 3: Comparison: ABP 710 vs Infliximab; The response difference at week 14 was estimated by the Mantel-Haenszel estimate; 90% confidence intervals were estimated from the stratified Newcombe confidence limits, adjusting for actual stratification factors (geographic region and prior biologic use); Test type: Other; Response Difference = 9.37, 90% CI 2-sided [-0.51 to 12.87]

3. Secondary Outcome: Percentage of Participants With an ACR20 Response After Week 22
Description: as for outcome 2
Time Frame: Baseline and weeks 30, 34, 38, 46, and 50
Population: Participants re-randomized at week 22 (includes participants initially randomized to ABP 710 who continued treatment with ABP 710 at week 22); participants with missing data at a given visit were counted as non-responders.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | ABP 710 / ABP 710 | Infliximab / Infliximab | Infliximab / ABP 710
Number analyzed (Participants) | 244 | 121 | 119
percentage of participants
  Week 30 | 69.7 [63.90 to 75.44] | 66.9 [58.56 to 75.32] | 74.8 [66.99 to 82.59]
  Week 34 | 74.6 [69.13 to 80.05] | 71.1 [63.00 to 79.15] | 74.8 [66.99 to 82.59]
  Week 38 | 70.5 [64.77 to 76.21] | 69.4 [61.21 to 77.63] | 72.3 [64.23 to 80.31]
  Week 46 | 61.9 [55.79 to 67.98] | 65.3 [56.81 to 73.77] | 66.4 [57.90 to 74.87]
  Week 50 | 67.6 [61.75 to 73.49] | 72.7 [64.79 to 80.66] | 70.6 [62.40 to 78.77]
Statistical Analysis 1: Comparison: ABP 710 / ABP 710 vs Infliximab / Infliximab; The response difference (ABP 710/ABP 710 minus Infliximab/Infliximab) at week 30 was estimated by the Mantel-Haenszel estimate; 90% confidence intervals were estimated from the stratified Newcombe confidence limits, adjusting for actual stratification factors (geographic region and prior biologic use); Test type: Other; Response Difference = 3.05, 90% CI 2-sided [-5.26 to 11.73]
Statistical Analysis 2: Comparison: Infliximab / Infliximab vs Infliximab / ABP 710; The response difference (Infliximab/ABP 710 minus Infliximab/Infliximab) at week 30 was estimated by the Mantel-Haenszel estimate; 90% confidence intervals were estimated from the stratified Newcombe confidence limits, adjusting for actual stratification factors (geographic region and prior biologic use); Test type: Other; Response Difference = 8.50, 90% CI 2-sided [-1.18 to 17.97]
Statistical Analysis 3: Comparison: ABP 710 / ABP 710 vs Infliximab / Infliximab; The response difference (ABP 710/ABP 710 minus Infliximab/Infliximab) at week 34 was estimated by the Mantel-Haenszel estimate; 90% confidence intervals were estimated from the stratified Newcombe confidence limits, adjusting for actual stratification factors (geographic region and prior biologic use); Test type: Other; Response Difference = 3.31, 90% CI 2-sided [-4.61 to 11.70]
Statistical Analysis 4: Comparison: Infliximab / Infliximab vs Infliximab / ABP 710; The response difference (Infliximab/ABP 710 minus Infliximab/Infliximab) at week 34 was estimated by the Mantel-Haenszel estimate; 90% confidence intervals were estimated from the stratified Newcombe confidence limits, adjusting for actual stratification factors (geographic region and prior biologic use); Test type: Other; Response Difference = 4.06, 90% CI 2-sided [-5.40 to 13.40]
Statistical Analysis 5: Comparison: ABP 710 / ABP 710 vs Infliximab / Infliximab; The response difference (ABP 710/ABP 710 minus Infliximab/Infliximab) at week 38 was estimated by the Mantel-Haenszel estimate; 90% confidence intervals were estimated from the stratified Newcombe confidence limits, adjusting for actual stratification factors (geographic region and prior biologic use); Test type: Other; Response Difference = 0.82, 90% CI 2-sided [-7.34 to 9.40]
Statistical Analysis 6: Comparison: Infliximab / Infliximab vs Infliximab / ABP 710; The response difference (Infliximab/ABP 710 minus Infliximab/Infliximab) at week 38 was estimated by the Mantel-Haenszel estimate; 90% confidence intervals were estimated from the stratified Newcombe confidence limits, adjusting for actual stratification factors (geographic region and prior biologic use); Test type: Other; Response Difference = 2.79, 90% CI 2-sided [-6.86 to 12.34]
Statistical Analysis 7: Comparison: ABP 710 / ABP 710 vs Infliximab / Infliximab; The response difference (ABP 710/ABP 710 minus Infliximab/Infliximab) at week 46 was estimated by the Mantel-Haenszel estimate; 90% confidence intervals were estimated from the stratified Newcombe confidence limits, adjusting for actual stratification factors (geographic region and prior biologic use); Test type: Other; Response Difference = -3.74, 90% CI 2-sided [-12.27 to 5.17]
Statistical Analysis 8: Comparison: Infliximab / Infliximab vs Infliximab / ABP 710; The response difference (Infliximab/ABP 710 minus Infliximab/Infliximab) at week 46 was estimated by the Mantel-Haenszel estimate; 90% confidence intervals were estimated from the stratified Newcombe confidence limits, adjusting for actual stratification factors (geographic region and prior biologic use); Test type: Other; Response Difference = 1.12, 90% CI 2-sided [-8.89 to 11.08]
Statistical Analysis 9: Comparison: ABP 710 / ABP 710 vs Infliximab / Infliximab; The response difference (ABP 710/ABP 710 minus Infliximab/Infliximab) at week 50 was estimated by the Mantel-Haenszel estimate; 90% confidence intervals were estimated from the stratified Newcombe confidence limits, adjusting for actual stratification factors (geographic region and prior biologic use); Test type: Other; Response Difference = -5.25, 90% CI 2-sided [-13.24 to 3.29]
Statistical Analysis 10: Comparison: Infliximab / Infliximab vs Infliximab / ABP 710; The response difference (Infliximab/ABP 710 minus Infliximab/Infliximab) at week 50 was estimated by the Mantel-Haenszel estimate; 90% confidence intervals were estimated from the stratified Newcombe confidence limits, adjusting for actual stratification factors (geographic region and prior biologic use); Test type: Other; Response Difference = -1.49, 90% CI 2-sided [-11.01 to 8.04]

4. Secondary Outcome: Percentage of Participants With an ACR50 Response Through Week 22
Description: A positive ACR50 response is defined if the following 3 criteria for improvement from baseline were met:
  * ≥ 50% improvement in 68 tender joint count;
  * ≥ 50% improvement in 66 swollen joint count; and
  * ≥ 50% improvement in at least 3 of the 5 following parameters:
    * Patient's assessment of disease-related pain (measured on a 100 mm visual analog scale [VAS]);
    * Patient's global health assessment (measured on a 100 mm VAS);
    * Investigator's global health assessment (measured on a 100 mm VAS);
    * Patient's self-assessment of physical function (Health Assessment Questionnaire - Disability Index [HAQ-DI]);
    * C-reactive protein concentration.
Time Frame: Baseline and weeks 2, 6, 14, and 22
Population: Intent-to-treat population; participants with missing data at a given visit were counted as non-responders.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | ABP 710 | Infliximab
Number analyzed (Participants) | 279 | 279
percentage of participants
  Week 2 | 17.2 [12.78 to 21.63] | 12.5 [8.66 to 16.43]
  Week 6 | 30.1 [24.72 to 35.49] | 28.3 [23.03 to 33.60]
  Week 14 | 39.4 [33.69 to 45.16] | 36.9 [31.25 to 42.58]
  Week 22 | 43.0 [37.20 to 48.82] | 36.2 [30.56 to 41.84]
Statistical Analysis 1: Comparison: ABP 710 vs Infliximab; [analysis description as in outcome 2, analysis 1]; Test type: Other; Response Difference = 4.41, 90% CI 2-sided [-0.56 to 9.38]
Statistical Analysis 2: Comparison: ABP 710 vs Infliximab; [analysis description as in outcome 2, analysis 2]; Test type: Other; Response Difference = 1.62, 90% CI 2-sided [-4.71 to 7.94]
Statistical Analysis 3: Comparison: ABP 710 vs Infliximab; [analysis description as in outcome 2, analysis 3]; Test type: Other; Response Difference = 2.30, 90% CI 2-sided [-4.45 to 9.03]
Statistical Analysis 4: Comparison: ABP 710 vs Infliximab; The response difference at week 22 was estimated by the Mantel-Haenszel estimate; 90% confidence intervals were estimated from the stratified Newcombe confidence limits, adjusting for actual stratification factors (geographic region and prior biologic use); Test type: Other; Response Difference = 7.09, 90% CI 2-sided [0.27 to 13.83]

5. Secondary Outcome: Percentage of Participants With an ACR50 Response After Week 22
Description: as for outcome 4
Time Frame: Baseline and weeks 30, 34, 38, 46, and 50
Population: as for outcome 3
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | ABP 710 / ABP 710 | Infliximab / Infliximab | Infliximab / ABP 710
Number analyzed (Participants) | 244 | 121 | 119
percentage of participants
  Week 30 | 43.0 [36.82 to 49.25] | 44.6 [35.77 to 53.49] | 47.1 [38.09 to 56.03]
  Week 34 | 52.5 [46.19 to 58.73] | 46.3 [37.40 to 55.17] | 56.3 [47.39 to 65.21]
  Week 38 | 48.0 [41.68 to 54.22] | 47.1 [38.21 to 56.00] | 49.6 [40.60 to 58.56]
  Week 46 | 43.9 [37.63 to 50.08] | 44.6 [35.77 to 53.49] | 50.4 [41.44 to 59.40]
  Week 50 | 49.2 [42.91 to 55.45] | 54.5 [45.67 to 63.42] | 57.1 [48.25 to 66.03]
Statistical Analysis 1: Comparison: ABP 710 / ABP 710 vs Infliximab / Infliximab; [analysis description as in outcome 3, analysis 1]; Test type: Other; Response Difference = -1.33, 90% CI 2-sided [-10.40 to 7.62]
Statistical Analysis 2: Comparison: Infliximab / Infliximab vs Infliximab / ABP 710; [analysis description as in outcome 3, analysis 2]; Test type: Other; Response Difference = 3.24, 90% CI 2-sided [-7.28 to 13.67]
Statistical Analysis 3: Comparison: ABP 710 / ABP 710 vs Infliximab / Infliximab; [analysis description as in outcome 3, analysis 3]; Test type: Other; Response Difference = 6.52, 90% CI 2-sided [-2.62 to 15.48]
Statistical Analysis 4: Comparison: Infliximab / Infliximab vs Infliximab / ABP 710; [analysis description as in outcome 3, analysis 4]; Test type: Other; Response Difference = 10.74, 90% CI 2-sided [0.12 to 21.03]
Statistical Analysis 5: Comparison: ABP 710 / ABP 710 vs Infliximab / Infliximab; [analysis description as in outcome 3, analysis 5]; Test type: Other; Response Difference = 0.56, 90% CI 2-sided [-8.54 to 9.59]
Statistical Analysis 6: Comparison: Infliximab / Infliximab vs Infliximab / ABP 710; [analysis description as in outcome 3, analysis 6]; Test type: Other; Response Difference = 2.93, 90% CI 2-sided [-7.62 to 13.39]
Statistical Analysis 7: Comparison: ABP 710 / ABP 710 vs Infliximab / Infliximab; [analysis description as in outcome 3, analysis 7]; Test type: Other; Response Difference = -1.04, 90% CI 2-sided [-10.11 to 7.93]
Statistical Analysis 8: Comparison: Infliximab / Infliximab vs Infliximab / ABP 710; [analysis description as in outcome 3, analysis 8]; Test type: Other; Response Difference = 6.14, 90% CI 2-sided [-4.44 to 16.54]
Statistical Analysis 9: Comparison: ABP 710 / ABP 710 vs Infliximab / Infliximab; [analysis description as in outcome 3, analysis 9]; Test type: Other; Response Difference = -5.43, 90% CI 2-sided [-14.39 to 3.71]
Statistical Analysis 10: Comparison: Infliximab / Infliximab vs Infliximab / ABP 710; [analysis description as in outcome 3, analysis 10]; Test type: Other; Response Difference = 2.98, 90% CI 2-sided [-7.51 to 13.37]

6. Secondary Outcome: Percentage of Participants With an ACR70 Response Through Week 22
Description: A positive ACR70 response is defined if the following 3 criteria for improvement from baseline were met:
  * ≥ 70% improvement in 68 tender joint count;
  * ≥ 70% improvement in 66 swollen joint count; and
  * ≥ 70% improvement in at least 3 of the 5 following parameters:
    * Patient's assessment of disease-related pain (measured on a 100 mm visual analog scale [VAS]);
    * Patient's global health assessment (measured on a 100 mm VAS);
    * Investigator's global health assessment (measured on a 100 mm VAS);
    * Patient's self-assessment of physical function (Health Assessment Questionnaire - Disability Index [HAQ-DI]);
    * C-reactive protein concentration.
Time Frame: Baseline and weeks 2, 6, 14, and 22
Population: Intent-to-treat population; participants with missing data at a given visit were counted as non-responders.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | ABP 710 | Infliximab
Number analyzed (Participants) | 279 | 279
percentage of participants
  Week 2 | 3.9 [1.66 to 6.23] | 6.5 [3.57 to 9.33]
  Week 6 | 14.3 [10.22 to 18.45] | 16.5 [12.13 to 20.84]
  Week 14 | 21.9 [17.01 to 26.71] | 16.1 [11.81 to 20.44]
  Week 22 | 24.0 [19.00 to 29.03] | 19.7 [15.05 to 24.38]
Statistical Analysis 1: Comparison: ABP 710 vs Infliximab; [analysis description as in outcome 2, analysis 1]; Test type: Other; Response Difference = -2.50, 90% CI 2-sided [-5.84 to 0.83]
Statistical Analysis 2: Comparison: ABP 710 vs Infliximab; [analysis description as in outcome 2, analysis 2]; Test type: Other; Response Difference = -2.43, 90% CI 2-sided [-7.47 to 2.64]
Statistical Analysis 3: Comparison: ABP 710 vs Infliximab; [analysis description as in outcome 2, analysis 3]; Test type: Other; Response Difference = 5.46, 90% CI 2-sided [-0.01 to 10.91]
Statistical Analysis 4: Comparison: ABP 710 vs Infliximab; [analysis description as in outcome 4, analysis 4]; Test type: Other; Response Difference = 4.58, 90% CI 2-sided [-1.21 to 10.34]

7. Secondary Outcome: Percentage of Participants With an ACR70 Response After Week 22
Description: as for outcome 6
Time Frame: Baseline and weeks 30, 34, 38, 46, and 50
Population: as for outcome 3
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | ABP 710 / ABP 710 | Infliximab / Infliximab | Infliximab / ABP 710
Number analyzed (Participants) | 244 | 121 | 119
percentage of participants
  Week 30 | 26.6 [21.09 to 32.19] | 26.4 [18.59 to 34.30] | 26.1 [18.16 to 33.94]
  Week 34 | 29.5 [23.79 to 35.23] | 28.1 [20.09 to 36.11] | 35.3 [26.71 to 43.88]
  Week 38 | 29.1 [23.40 to 34.80] | 29.8 [21.61 to 37.90] | 32.8 [24.34 to 41.21]
  Week 46 | 29.5 [23.79 to 35.23] | 29.8 [21.61 to 37.90] | 37.0 [28.30 to 45.65]
  Week 50 | 34.0 [28.07 to 39.96] | 32.2 [23.90 to 40.56] | 43.7 [34.79 to 52.61]
Statistical Analysis 1: Comparison: ABP 710 / ABP 710 vs Infliximab / Infliximab; [analysis description as in outcome 3, analysis 1]; Test type: Other; Response Difference = 0.20, 90% CI 2-sided [-8.12 to 8.02]
Statistical Analysis 2: Comparison: Infliximab / Infliximab vs Infliximab / ABP 710; [analysis description as in outcome 3, analysis 2]; Test type: Other; Response Difference = -0.08, 90% CI 2-sided [-9.39 to 9.28]
Statistical Analysis 3: Comparison: ABP 710 / ABP 710 vs Infliximab / Infliximab; [analysis description as in outcome 3, analysis 3]; Test type: Other; Response Difference = 1.50, 90% CI 2-sided [-7.00 to 9.51]
Statistical Analysis 4: Comparison: Infliximab / Infliximab vs Infliximab / ABP 710; [analysis description as in outcome 3, analysis 4]; Test type: Other; Response Difference = 7.49, 90% CI 2-sided [-2.39 to 17.22]
Statistical Analysis 5: Comparison: ABP 710 / ABP 710 vs Infliximab / Infliximab; [analysis description as in outcome 3, analysis 5]; Test type: Other; Response Difference = -0.50, 90% CI 2-sided [-9.03 to 7.59]
Statistical Analysis 6: Comparison: Infliximab / Infliximab vs Infliximab / ABP 710; [analysis description as in outcome 3, analysis 6]; Test type: Other; Response Difference = 3.39, 90% CI 2-sided [-6.41 to 13.14]
Statistical Analysis 7: Comparison: ABP 710 / ABP 710 vs Infliximab / Infliximab; [analysis description as in outcome 3, analysis 7]; Test type: Other; Response Difference = -0.43, 90% CI 2-sided [-8.98 to 7.66]
Statistical Analysis 8: Comparison: Infliximab / Infliximab vs Infliximab / ABP 710; [analysis description as in outcome 3, analysis 8]; Test type: Other; Response Difference = 7.87, 90% CI 2-sided [-2.13 to 17.68]
Statistical Analysis 9: Comparison: ABP 710 / ABP 710 vs Infliximab / Infliximab; [analysis description as in outcome 3, analysis 9]; Test type: Other; Response Difference = 1.95, 90% CI 2-sided [-6.81 to 10.29]
Statistical Analysis 10: Comparison: Infliximab / Infliximab vs Infliximab / ABP 710; [analysis description as in outcome 3, analysis 10]; Test type: Other; Response Difference = 12.06, 90% CI 2-sided [1.74 to 22.04]

8. Secondary Outcome: Change From Baseline in Disease Activity Score 28 (DAS28) Through Week 22
Description: The DAS28 measures the severity of disease at a specific time and is derived from the following variables:
  * 28 tender joint count
  * 28 swollen joint count
  * C-reactive protein (CRP)
  * Patient's global health assessment measured on a 100 mm VAS, where 0 mm = no RA activity and 100 mm = worst RA activity imaginable.
  DAS28(CRP) scores range from 0 to approximately 10, with the upper bound dependent on the highest possible level of CRP. A DAS28 score higher than 5.1 indicates high disease activity, a DAS28 score less than 3.2 indicates low disease activity, and a DAS28 score less than 2.6 indicates clinical remission.
Time Frame: Baseline and weeks 2, 6, 14, and 22
Population: Intent-to-treat population with available data at each time point.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | ABP 710 | Infliximab
Number analyzed (Participants) | 279 | 279
units on a scale
  Week 2: number analyzed (Participants) | 260 | 255
  Week 2 | -1.36 (0.991) | -1.29 (1.006)
  Week 6: number analyzed (Participants) | 259 | 253
  Week 6 | -1.82 (1.222) | -1.82 (1.203)
  Week 14: number analyzed (Participants) | 253 | 250
  Week 14 | -1.95 (1.218) | -1.91 (1.289)
  Week 22: number analyzed (Participants) | 245 | 243
  Week 22 | -2.06 (1.290) | -2.06 (1.296)
Statistical Analysis 1: Comparison: ABP 710 vs Infliximab; Week 2 difference between means (ABP 710 minus infliximab) and 90% CIs for difference between means were based on ANCOVA model with the DAS28-CRP change from baseline as the response and adjusted for the baseline DAS28-CRP measurement and the actual stratification factors: geographic region and prior biologic use for RA; Test type: Other; Mean Difference = -0.07, 90% CI 2-sided [-0.20 to 0.007]
Statistical Analysis 2: Comparison: ABP 710 vs Infliximab; Week 6 difference between means (ABP 710 minus infliximab) and 90% CIs for difference between means were based on ANCOVA model with the DAS28-CRP change from baseline as the response and adjusted for the baseline DAS28-CRP measurement and the actual stratification factors: geographic region and prior biologic use for RA; Test type: Other; Mean Difference = 0.00, 90% CI 2-sided [-0.17 to 0.16]
Statistical Analysis 3: Comparison: ABP 710 vs Infliximab; Week 14 difference between means (ABP 710 minus infliximab) and 90% CIs for difference between means were based on ANCOVA model with the DAS28-CRP change from baseline as the response and adjusted for the baseline DAS28-CRP measurement and the actual stratification factors: geographic region and prior biologic use for RA; Test type: Other; Mean Difference = -0.04, 90% CI 2-sided [-0.21 to 0.14]
Statistical Analysis 4: Comparison: ABP 710 vs Infliximab; Week 22 difference between means (ABP 710 minus infliximab) and 90% CIs for difference between means were based on ANCOVA model with the DAS28-CRP change from baseline as the response and adjusted for the baseline DAS28-CRP measurement and the actual stratification factors: geographic region and prior biologic use for RA; Test type: Other; Mean Difference = -0.01, 90% CI 2-sided [-0.20 to 0.17]

9. Secondary Outcome: Change From Baseline in Disease Activity Score 28 (DAS28) After Week 22
Description: as for outcome 8
Time Frame: Baseline and weeks 30, 34, 38, 46, and 50
Population: Participants re-randomized at week 22 (includes participants initially randomized to ABP 710 who continued treatment with ABP 710 at week 22) and with available data at each time point.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | ABP 710 / ABP 710 | Infliximab / Infliximab | Infliximab / ABP 710
Number analyzed (Participants) | 244 | 121 | 119
units on a scale
  Week 30: number analyzed (Participants) | 225 | 112 | 112
  Week 30 | -2.07 (1.278) | -2.25 (1.379) | -2.22 (1.266)
  Week 34: number analyzed (Participants) | 222 | 113 | 111
  Week 34 | -2.32 (1.306) | -2.46 (1.372) | -2.45 (1.309)
  Week 38: number analyzed (Participants) | 219 | 114 | 110
  Week 38 | -2.20 (1.277) | -2.27 (1.301) | -2.32 (1.400)
  Week 46: number analyzed (Participants) | 205 | 108 | 108
  Week 46 | -2.11 (1.381) | -2.27 (1.387) | -2.26 (1.440)
  Week 50: number analyzed (Participants) | 203 | 110 | 107
  Week 50 | -2.45 (1.365) | -2.49 (1.276) | -2.64 (1.328)
Statistical Analysis 1: Comparison: ABP 710 / ABP 710 vs Infliximab / Infliximab; Week 30 difference between means (ABP 710/ABP 710 minus Infliximab/Infliximab) and 90% CIs for difference between means were based on ANCOVA model with the DAS28-CRP change from baseline as the response and adjusted for the baseline DAS28-CRP measurement and the actual stratification factors: geographic region and prior biologic use for RA; Test type: Other; Mean Difference = 0.16, 90% CI 2-sided [-0.08 to 0.40]
Statistical Analysis 2: Comparison: Infliximab / Infliximab vs Infliximab / ABP 710; Week 30 difference between means (Infliximab/ABP 710 minus Infliximab/Infliximab) and 90% CIs for difference between means were based on ANCOVA model with the DAS28-CRP change from baseline as the response and adjusted for the baseline DAS28-CRP measurement and the actual stratification factors: geographic region and prior biologic use for RA; Test type: Other; Mean Difference = 0.00, 90% CI 2-sided [-0.27 to 0.28]
Statistical Analysis 3: Comparison: ABP 710 / ABP 710 vs Infliximab / Infliximab; Week 34 difference between means (ABP 710/ABP 710 minus Infliximab/Infliximab) and 90% CIs for difference between means were based on ANCOVA model with the DAS28-CRP change from baseline as the response and adjusted for the baseline DAS28-CRP measurement and the actual stratification factors: geographic region and prior biologic use for RA; Test type: Other; Mean Difference = 0.11, 90% CI 2-sided [-0.12 to 0.35]
Statistical Analysis 4: Comparison: Infliximab / Infliximab vs Infliximab / ABP 710; Week 34 difference between means (Infliximab/ABP 710 minus Infliximab/Infliximab) and 90% CIs for difference between means were based on ANCOVA model with the DAS28-CRP change from baseline as the response and adjusted for the baseline DAS28-CRP measurement and the actual stratification factors: geographic region and prior biologic use for RA; Test type: Other; Mean Difference = -0.03, 90% CI 2-sided [-0.30 to 0.24]
Statistical Analysis 5: Comparison: ABP 710 / ABP 710 vs Infliximab / Infliximab; Week 38 difference between means (ABP 710/ABP 710 minus Infliximab/Infliximab) and 90% CIs for difference between means were based on ANCOVA model with the DAS28-CRP change from baseline as the response and adjusted for the baseline DAS28-CRP measurement and the actual stratification factors: geographic region and prior biologic use for RA; Test type: Other; Mean Difference = 0.06, 90% CI 2-sided [-0.18 to 0.30]
Statistical Analysis 6: Comparison: Infliximab / Infliximab vs Infliximab / ABP 710; Week 38 difference between means (Infliximab/ABP 710 minus Infliximab/Infliximab) and 90% CIs for difference between means were based on ANCOVA model with the DAS28-CRP change from baseline as the response and adjusted for the baseline DAS28-CRP measurement and the actual stratification factors: geographic region and prior biologic use for RA; Test type: Other; Mean Difference = -0.08, 90% CI 2-sided [-0.36 to 0.20]
Statistical Analysis 7: Comparison: ABP 710 / ABP 710 vs Infliximab / Infliximab; Week 46 difference between means (ABP 710/ABP 710 minus Infliximab/Infliximab) and 90% CIs for difference between means were based on ANCOVA model with the DAS28-CRP change from baseline as the response and adjusted for the baseline DAS28-CRP measurement and the actual stratification factors: geographic region and prior biologic use for RA; Test type: Other; Mean Difference = 0.11, 90% CI 2-sided [-0.14 to 0.37]
Statistical Analysis 8: Comparison: Infliximab / Infliximab vs Infliximab / ABP 710; Week 46 difference between means (Infliximab/ABP 710 minus Infliximab/Infliximab) and 90% CIs for difference between means were based on ANCOVA model with the DAS28-CRP change from baseline as the response and adjusted for the baseline DAS28-CRP measurement and the actual stratification factors: geographic region and prior biologic use for RA; Test type: Other; Mean Difference = -0.05, 90% CI 2-sided [-0.34 to 0.25]
Statistical Analysis 9: Comparison: ABP 710 / ABP 710 vs Infliximab / Infliximab; Week 50 difference between means (ABP 710/ABP 710 minus Infliximab/Infliximab) and 90% CIs for difference between means were based on ANCOVA model with the DAS28-CRP change from baseline as the response and adjusted for the baseline DAS28-CRP measurement and the actual stratification factors: geographic region and prior biologic use for RA; Test type: Other; Mean Difference = 0.00, 90% CI 2-sided [-0.24 to 0.24]
Statistical Analysis 10: Comparison: Infliximab / Infliximab vs Infliximab / ABP 710; Week 50 difference between means (Infliximab/ABP 710 minus Infliximab/Infliximab) and 90% CIs for difference between means were based on ANCOVA model with the DAS28-CRP change from baseline as the response and adjusted for the baseline DAS28-CRP measurement and the actual stratification factors: geographic region and prior biologic use for RA; Test type: Other; Mean Difference = -0.20, 90% CI 2-sided [-0.47 to 0.08]

ADVERSE EVENTS:
Time Frame: From first dose to week 22 (initial ABP 710 and infliximab treatment groups) and from week 22 to week 50 for participants re-randomized at week 22, or up to 28 days after last dose for participants who discontinued early.
Description: Other Adverse Events summarizes the non-serious occurrences of adverse events that exceed the indicated frequency threshold.
Groups:
- ABP 710: Participants received 3 mg/kg intravenous (IV) infusion of ABP 710 on day 1, at weeks 2 and 6, and every 8 weeks thereafter until week 22.
- Infliximab: Participants received 3 mg/kg IV infusion of infliximab on day 1, at weeks 2 and 6, and every 8 weeks thereafter until week 22.
Arm/Group | ABP 710 | Infliximab | ABP 710 / ABP 710 | Infliximab / Infliximab | Infliximab / ABP 710
All-Cause Mortality (participants affected / at risk) | 1/278 | 1/278 | 0/241 | 0/121 | 0/119
Serious Adverse Events (participants affected / at risk) | 9/278 | 14/278 | 15/241 | 4/121 | 1/119
Other Adverse Events (participants affected / at risk) | 48/278 | 32/278 | 52/241 | 28/121 | 30/119
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | ABP 710 (N=278) | Infliximab (N=278) | ABP 710 / ABP 710 (N=241) | Infliximab / Infliximab (N=121) | Infliximab / ABP 710 (N=119)
Iron deficiency anaemia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 1
Microcytic anaemia (Blood and lymphatic system disorders) | 0 | 0 | 1 | 0 | 0
Acute myocardial infarction (Cardiac disorders) | 0 | 1 | 0 | 0 | 0
Cardiac failure congestive (Cardiac disorders) | 0 | 0 | 1 | 0 | 0
Cardiovascular insufficiency (Cardiac disorders) | 1 | 0 | 0 | 0 | 0
Myocardial infarction (Cardiac disorders) | 0 | 1 | 0 | 0 | 0
Ventricular extrasystoles (Cardiac disorders) | 1 | 0 | 0 | 0 | 0
Colitis (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0
Constipation (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0
Pancreatitis acute (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0
Chest discomfort (General disorders) | 1 | 0 | 0 | 0 | 0
Non-cardiac chest pain (General disorders) | 0 | 0 | 1 | 0 | 0
Jaundice cholestatic (Hepatobiliary disorders) | 0 | 0 | 0 | 1 | 0
Appendicitis (Infections and infestations) | 0 | 0 | 1 | 0 | 0
Arthritis bacterial (Infections and infestations) | 0 | 1 | 0 | 0 | 0
Cellulitis (Infections and infestations) | 0 | 0 | 2 | 0 | 0
Febrile infection (Infections and infestations) | 1 | 0 | 0 | 0 | 0
Gastroenteritis (Infections and infestations) | 0 | 0 | 1 | 0 | 0
Pneumonia bacterial (Infections and infestations) | 0 | 1 | 0 | 0 | 0
Pneumonia legionella (Infections and infestations) | 0 | 1 | 0 | 0 | 0
Pneumonia pneumococcal (Infections and infestations) | 1 | 0 | 0 | 0 | 0
Pneumonia viral (Infections and infestations) | 0 | 1 | 0 | 0 | 0
Femoral neck fracture (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0 | 0
Hip fracture (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0 | 0
Laceration (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0 | 0
Multiple injuries (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0 | 0
Tibia fracture (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0 | 0
Transaminases increased (Investigations) | 0 | 0 | 1 | 0 | 0
Dehydration (Metabolism and nutrition disorders) | 0 | 0 | 1 | 0 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1 | 0
Foot deformity (Musculoskeletal and connective tissue disorders) | 0 | 0 | 2 | 0 | 0
Muscular weakness (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0 | 0
Rheumatoid arthritis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 1
Chronic lymphocytic leukaemia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 0 | 0
Endometrial adenocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 0 | 0
Malignant melanoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1 | 0 | 0
Ovarian low malignant potential tumour (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 0 | 0
Transitional cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 0 | 0
Sciatica (Nervous system disorders) | 1 | 0 | 0 | 0 | 0
Transient ischaemic attack (Nervous system disorders) | 1 | 0 | 0 | 0 | 0
Nephrolithiasis (Renal and urinary disorders) | 0 | 1 | 0 | 0 | 0
Renal failure (Renal and urinary disorders) | 0 | 1 | 0 | 0 | 0
Ureterolithiasis (Renal and urinary disorders) | 0 | 1 | 0 | 0 | 0
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1 | 0
Dermatitis atopic (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1 | 0
Orthostatic hypotension (Vascular disorders) | 0 | 1 | 0 | 0 | 0
Peripheral ischaemia (Vascular disorders) | 0 | 0 | 1 | 0 | 0
Thrombosis (Vascular disorders) | 0 | 2 | 0 | 0 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | ABP 710 (N=278) | Infliximab (N=278) | ABP 710 / ABP 710 (N=241) | Infliximab / Infliximab (N=121) | Infliximab / ABP 710 (N=119)
Nasopharyngitis (Infections and infestations) | 12 | 4 | 13 | 11 | 8
Pharyngitis (Infections and infestations) | 8 | 3 | 2 | 2 | 7
Upper respiratory tract infection (Infections and infestations) | 17 | 18 | 23 | 9 | 14
Rheumatoid arthritis (Musculoskeletal and connective tissue disorders) | 14 | 11 | 23 | 9 | 7

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Clinical Trial Agreement generally does not restrict an investigator's discussion of trial results after completion. The Agreement permits Amgen a limited period of time to review material discussing trial results (typically up to 45 days and possible extension). Amgen may remove confidential information, but authors have final control and approval of publication content. For multicenter studies, the investigator agrees not to publish any results before the first multi-center publication.

DOCUMENTS (2):
  • Study Protocol (2017-03-17): https://cdn.clinicaltrials.gov/large-docs/01/NCT02937701/Prot_000.pdf
  • Statistical Analysis Plan (2018-06-06): https://cdn.clinicaltrials.gov/large-docs/01/NCT02937701/SAP_001.pdf